CLINICAL TRIAL: NCT05462990
Title: A Randomized, Two-arm, Placebo-controlled, Participant, Investigator and Sponsor-blinded, Proof-of-concept Study Investigating the Efficacy, Safety and Tolerability of QUC398 in Patients With Symptomatic Knee Osteoarthritis
Brief Title: A Proof-of-concept Study to Examine QUC398 in Participants With Knee OA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CQUC398A12201; 2021-002795-39 (EudraCT Number); 2023-509274-28-00 (Other: EU CT)
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Osteoarthritis, Knee
Keywords: QUC398; Osteoarthritis of Knee; Osteoarthritis of the Knee; Knee joint; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: participant, investigator and sponsor-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- QUC398 300 mg (Experimental): QUC398 was administered subcutaneous every 4 weeks during 48 weeks.
  Interventions: Drug: QUC398
- Placebo (Placebo Comparator): Placebo was administered subcutaneous every 4 weeks during 48 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QUC398 — QUC398 150 mg/mL, solution for subcutaneous (s.c) injection (1 mL). 2 injections were administered to complete 300 mg.
  Arms: QUC398 300 mg
Drug: Placebo — Matching Placebo solution for s.c. injection (1 mL). 2 injections were administered per dose to ensure blinding.
  Arms: Placebo

SUMMARY:
The purpose of the study was to find out if the investigational treatment named QUC398 had beneficial effects on osteoarthritis (OA) knee pain and knee cartilage, and if it was safe and tolerated.

DETAILED DESCRIPTION:
This was a non-confirmatory study using a randomized, placebo-controlled, parallel-group, participant, investigator and sponsor-blinded design to investigate efficacy, safety and tolerability of subcutaneous injections of QUC398 300 mg vs placebo every 4 weeks (q4w) in participants with symptomatic knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Weight ≥ 50 kg and body mass index 18 -35 kg/m2 at Screening 1
* Kellgren-Lawrence grade 2 to 4 in the tibio-femoral compartment in the target knee confirmed by radiography in standing weight-bearing fixed flexion position and posterior-anterior view, at Screening 1
* mJSN 1-2 in the medial tibiofemoral compartment of the target knee, confirmed with Xray by central reader at Screening 1
* Symptomatic OA with moderate to severe pain (corresponding to Pain NRS ≥ 5 to ≤ 9) in the target knee for the majority of days in the last 3 months prior to Screening 1, as per participant's judgement
* Symptomatic OA with moderate to severe pain (corresponding to Pain NRS ≥ 5 to ≤ 9) in the target knee at Screening 1 and 2
* Moderate to severe OA pain (corresponding to Pain NRS ≥5 to ≤9) in the target knee during the last 7 days prior to Screening 3, confirmed by:

Completed pain diary for at least 6 of the last 7 days prior to Screening 3, AND Diary reported Pain NRS ≥5 to ≤9 for at least 6 of the last 7 days prior to Screening 3

- KOOS pain subscale ≤ 60 in the target knee at Screening 1, Screening 2, and Screening 3

Exclusion Criteria:

* Painful ipsilateral hip OA defined as a Pain NRS ≥3 on the majority of days in the last 3 months prior to Screening 1, as reported by the patient
* Symptomatic, patello-femoral pain in the target knee as per investigator's examination at Screening 1
* Severe malalignment > 7.5º in the target knee (either varus or valgus), measured using standardized knee X-ray at Screening 1
* Patient unable or unwilling to undergo MRI or presenting absolute contraindications to MRI
* Previous exposure to any ADAMTS-5 drug, including QUC398.
* History or current diagnosis of ECG abnormalities

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2025-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- United States (3):
  - Clinical Research of West Florida Inc, Tampa, Florida
  - Boston Univ School of Medicine, Boston, Massachusetts
  - West Clinical Research, Morehead City, North Carolina
- Australia (3):
  - Novartis Investigative Site, Southport, Queensland
  - Novartis Investigative Site, Christchurch
  - Novartis Investigative Site, St Leonards
- Denmark (2):
  - Novartis Investigative Site, Herlev
  - Novartis Investigative Site, Vejle
- France (2):
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Orléans
- Spain (4):
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Leganés, Madrid
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Seville

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 14 investigative sites in 6 countries.
Pre-assignment Details: The study consisted of a screening period of up to approximately 6 weeks.
Period: Overall Study
Arm/Group | QUC398 300 mg | Placebo
Started | 50 | 51
Completed | 26 | 26
Not Completed | 24 | 25
Not completed — Adverse Event | 3 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Deviation | 3 | 1
Not completed — Study Terminated By Sponsor | 14 | 18
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QUC398 300 mg | Placebo | Total
Number analyzed (Participants) | 50 | 51 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (7.81) | 62.3 (7.10) | 64.1 (7.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 30 | 58
  Male | 22 | 21 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 48 | 49 | 97
  Black or African American | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain Subscale at Week 12
Description: The KOOS questionnaire is a commonly used instrument to assess the patient's perception about their knee and associated problems. The original KOOS consists of 5 subscales. One of those is the pain frequency/severity during functional activities consisting of 9 questions with a recall of 7 days. Each question has 5 standardized answer options with a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. Change from baseline in KOOS pain score was analyzed using a mixed effects model for repeated measures (MMRM) including all time-points to compare treatment groups. The model includes baseline, treatment, timepoint and treatment-by-timepoints as fixed effects. Missing data is assumed to be Missing at Random (MAR). Based on a primary estimand framework.
Time Frame: Baseline, Week 12
Population: The full analysis set (FAS) included all participants that received any study drug. Only participants with non-missing values were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | QUC398 300 mg | Placebo
Number analyzed (Participants) | 41 | 43
score on scale | 9.0 (2.25) | 17.5 (2.17)
Statistical Analysis 1: Comparison: QUC398 300 mg vs Placebo; Test type: Superiority; p = 0.9961, Mixed effects model for repeated measure — 1-sided p-value; Least Square Mean = -8.5249, 90% CI 2-sided [-13.7 to -3.3], Standard Error of Mean 3.1275

2. Secondary Outcome: Change From Baseline in Cartilage Volume of the Knee Index Region Measured by 3D-MRI
Description: Magnetic resonance images (MRI) were obtained from the target knee to visualize and quantify changes in volume of cartilage in the index region. The index region was defined as the union of the femoral medial anterior (FMA), central (FMC) and posterior (FMP) cartilage subregions in the knee. Change from baseline in cartilage volume was analyzed using a mixed effects model for repeated measures (MMRM) including all time-points to compare treatment groups. The model includes baseline, treatment, timepoint and treatment-timepoints as fixed effects, and participant as random effect. Missing data is assumed to be Missing at Random (MAR). Based on a secondary estimand framework.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm^3
Arm/Group | QUC398 300 mg | Placebo
Number analyzed (Participants) | 24 | 22
mm^3 | 47.8 (46.02) | 15.1 (47.42)

3. Secondary Outcome: Change From Baseline in Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain Subscale
Description: The KOOS questionnaire is a commonly used instrument to assess the patient's perception about their knee and associated problems. The original KOOS consists of 5 subscales. One of those is the pain frequency/severity during functional activities consisting of 9 questions with a recall of 7 days. Each question has 5 standardized answer options with a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. A positive change from baseline indicates an improvement. Change from baseline in KOOS pain score was analyzed using a mixed effects model for repeated measures (MMRM) including all time-points to compare treatment groups. The model includes baseline, treatment, timepoint and treatment-by-timepoints as fixed effects. Missing data is assumed to be Missing at Random (MAR). Based on second secondary estimand framework.
Time Frame: Baseline, Weeks 1 (Day 5), 4, 8, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: The full analysis set (FAS) included all participants that received any study drug. At each time point, only participants with non-missing values were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | QUC398 300 mg | Placebo
Number analyzed (Participants) | 45 | 49
score on scale
  Week 1 (Day 5) | 1.4 (1.17) | 5.0 (1.12)
  Week 4: number analyzed (Participants) | 43 | 48
  Week 4 | 3.9 (1.76) | 9.0 (1.67)
  Week 8: number analyzed (Participants) | 41 | 44
  Week 8 | 7.5 (1.88) | 14.1 (1.81)
  Week 16: number analyzed (Participants) | 43 | 47
  Week 16 | 11.8 (2.36) | 18.4 (2.28)
  Week 20: number analyzed (Participants) | 41 | 45
  Week 20 | 12.7 (2.3) | 18.1 (2.22)
  Week 24: number analyzed (Participants) | 38 | 45
  Week 24 | 11.8 (2.62) | 19.1 (2.5)
  Week 28: number analyzed (Participants) | 37 | 44
  Week 28 | 12.6 (2.64) | 21.2 (2.51)
  Week 32: number analyzed (Participants) | 36 | 44
  Week 32 | 10.9 (2.77) | 20.4 (2.61)
  Week 36: number analyzed (Participants) | 33 | 37
  Week 36 | 11.3 (2.74) | 21.7 (2.62)
  Week 40: number analyzed (Participants) | 29 | 29
  Week 40 | 12.9 (2.98) | 20.0 (2.92)
  Week 44: number analyzed (Participants) | 26 | 27
  Week 44 | 14.2 (3.33) | 19.0 (3.26)
  Week 48: number analyzed (Participants) | 23 | 23
  Week 48 | 11.7 (2.93) | 21.4 (2.87)
  Week 52: number analyzed (Participants) | 25 | 23
  Week 52 | 11.7 (2.95) | 20.8 (2.93)

4. Secondary Outcome: Change From Baseline in Pain Assessed by a Pain Numerical Rating Scale (NRS)
Description: The Numerical Rating Scale (NRS) Pain is a subjective assessment in which individuals rate their pain on an eleven-point numerical scale. NRS pain score ranges from 0-10 and for analyses were transformed to a 0-100 scale to be consistent with KOOS pain scores. A negative change from baseline implied improvement in pain. The NRS Pain instrument had a recall period of 24 hours and the participants were asked to rate the pain intensity at its worst. Change from baseline in NRS pain score was analyzed using a MMRM including all time-points to compare treatment groups. The model includes baseline, treatment, timepoint and treatment-by-timepoints as fixed effects. Missing data is assumed to be Missing at Random (MAR). Based on second secondary estimand framework.
Time Frame: Baseline, Weeks 1 (Day 5), 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | QUC398 300 mg | Placebo
Number analyzed (Participants) | 45 | 49
score on scale
  Week 1 (Day 5) | -2.6 (2.94) | -3.1 (2.83)
  Week 4: number analyzed (Participants) | 43 | 48
  Week 4 | -3.8 (2.97) | -8.7 (2.84)
  Week 8: number analyzed (Participants) | 41 | 44
  Week 8 | -7.5 (3.00) | -12.5 (2.88)
  Week 12: number analyzed (Participants) | 43 | 44
  Week 12 | -8.5 (2.98) | -18.1 (2.89)
  Week 16: number analyzed (Participants) | 43 | 47
  Week 16 | -12.8 (2.98) | -19.4 (2.86)
  Week 20: number analyzed (Participants) | 41 | 45
  Week 20 | -13.4 (3.01) | -17.9 (2.89)
  Week 24: number analyzed (Participants) | 38 | 45
  Week 24 | -10.7 (3.07) | -19.0 (2.90)
  Week 28: number analyzed (Participants) | 37 | 44
  Week 28 | -13.1 (3.10) | -23.5 (2.92)
  Week 32: number analyzed (Participants) | 36 | 43
  Week 32 | -13.6 (3.14) | -21.0 (2.95)
  Week 36: number analyzed (Participants) | 33 | 37
  Week 36 | -15.7 (3.22) | -23.5 (3.06)
  Week 40: number analyzed (Participants) | 29 | 29
  Week 40 | -16.4 (3.36) | -23.7 (3.28)
  Week 44: number analyzed (Participants) | 26 | 27
  Week 44 | -16.6 (3.48) | -21.3 (3.40)
  Week 48: number analyzed (Participants) | 23 | 23
  Week 48 | -15.6 (3.63) | -25.7 (3.59)
  Week 52: number analyzed (Participants) | 25 | 23
  Week 52 | -16.7 (3.61) | -25.4 (3.65)

5. Secondary Outcome: Change From Baseline in Total Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: The KOOS questionnaire is a commonly used instrument to assess the patient's perception about their knee and associated problems.The original KOOS consists of 5 subscales: Pain, other Symptoms (like stiffness and swelling), Function in Daily Living, Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL). A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. Total KOOS scale was calculated as the average of all subscales (100 indicating no symptoms and 0 indicating extreme symptoms). A positive change from baseline indicates an improvement. Change from baseline in KOOS total score was analyzed using a mixed effects model for repeated measures (MMRM) including all time-points to compare treatment groups. The model includes baseline, treatment, timepoint and treatment-by-timepoints as fixed effects. Missing data is assumed to be Missing at Random (MAR). Based on second secondary estimand framework.
Time Frame: Baseline, Weeks 1 (Day 5), 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | QUC398 300 mg | Placebo
Number analyzed (Participants) | 45 | 49
score on scale
  Week 1 (Day 5) | 1.4 (2.07) | 4.2 (1.99)
  Week 4: number analyzed (Participants) | 43 | 48
  Week 4 | 3.3 (2.08) | 8.4 (1.99)
  Week 8: number analyzed (Participants) | 41 | 44
  Week 8 | 6.7 (2.10) | 12.5 (2.02)
  Week 12: number analyzed (Participants) | 43 | 44
  Week 12 | 8.6 (2.09) | 15.9 (2.02)
  Week 16: number analyzed (Participants) | 43 | 47
  Week 16 | 10.8 (2.09) | 16.5 (2.01)
  Week 20: number analyzed (Participants) | 41 | 45
  Week 20 | 11.2 (2.11) | 16.2 (2.02)
  Week 24: number analyzed (Participants) | 38 | 45
  Week 24 | 10.6 (2.13) | 17.9 (2.03)
  Week 28: number analyzed (Participants) | 37 | 44
  Week 28 | 11.1 (2.16) | 19.2 (2.04)
  Week 32: number analyzed (Participants) | 36 | 44
  Week 32 | 11.1 (2.18) | 18.4 (2.05)
  Week 36: number analyzed (Participants) | 33 | 37
  Week 36 | 11.6 (2.23) | 20.1 (2.12)
  Week 40: number analyzed (Participants) | 29 | 29
  Week 40 | 12.7 (2.30) | 19.6 (2.24)
  Week 44: number analyzed (Participants) | 26 | 27
  Week 44 | 12.9 (2.38) | 18.4 (2.32)
  Week 48: number analyzed (Participants) | 23 | 23
  Week 48 | 12.5 (2.49) | 22.6 (2.46)
  Week 52: number analyzed (Participants) | 25 | 23
  Week 52 | 13.7 (2.49) | 21.0 (2.51)

6. Secondary Outcome: Change From Baseline in Knee Injury and Osteoarthritis Outcome Score (KOOS) Other Symptoms Subscale
Description: The KOOS questionnaire is a commonly used instrument to assess the patient's perception about their knee and associated problems. The original KOOS consists of 5 subscales. One of those is other symptoms (eg., stiffness, swelling, clicking) consisting of 7 questions with a recall of 7 days. Each question has 5 standardized answer options with a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. A positive change from baseline indicates an improvement. Change from baseline in KOOS Other symptoms score was analyzed using a mixed effects model for repeated measures (MMRM) including all time-points to compare treatment groups. The model includes baseline, treatment, timepoint and treatment-by-timepoints as fixed effects. Missing data is assumed to be Missing at Random (MAR). Based on second secondary estimand framework.
Time Frame: Baseline, Weeks 1 (Day 5), 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | QUC398 300 mg | Placebo
Number analyzed (Participants) | 45 | 49
score on scale
  Week 1 (Day 5) | 0.3 (2.23) | 4 (2.14)
  Week 4: number analyzed (Participants) | 43 | 48
  Week 4 | 2.5 (2.24) | 8.8 (2.15)
  Week 8: number analyzed (Participants) | 41 | 44
  Week 8 | 3.2 (2.26) | 12.3 (2.17)
  Week 12: number analyzed (Participants) | 43 | 44
  Week 12 | 6.6 (2.24) | 14.3 (2.18)
  Week 16: number analyzed (Participants) | 43 | 47
  Week 16 | 9.2 (2.24) | 15.5 (2.16)
  Week 20: number analyzed (Participants) | 41 | 45
  Week 20 | 8.7 (2.27) | 13.4 (2.18)
  Week 24: number analyzed (Participants) | 38 | 45
  Week 24 | 7.7 (2.3) | 14.6 (2.18)
  Week 28: number analyzed (Participants) | 37 | 44
  Week 28 | 7.6 (2.32) | 17.7 (2.2)
  Week 32: number analyzed (Participants) | 36 | 44
  Week 32 | 7.4 (2.35) | 15.7 (2.2)
  Week 36: number analyzed (Participants) | 33 | 37
  Week 36 | 8.2 (2.4) | 18.3 (2.28)
  Week 40: number analyzed (Participants) | 29 | 29
  Week 40 | 10.4 (2.48) | 16.9 (2.43)
  Week 44: number analyzed (Participants) | 26 | 27
  Week 44 | 11.1 (2.57) | 14.1 (2.51)
  Week 48: number analyzed (Participants) | 23 | 23
  Week 48 | 9.5 (2.68) | 18.6 (2.65)
  Week 52: number analyzed (Participants) | 25 | 23
  Week 52 | 11.1 (2.68) | 18.1 (2.7)

7. Secondary Outcome: Change From Baseline in Knee Injury and Osteoarthritis Outcome Score (KOOS) Function in Daily Living Subscale
Description: The KOOS questionnaire is a commonly used instrument to assess the patient's perception about their knee and associated problems. The original KOOS consists of 5 subscales. One of those is the Function in Daily Living consisting of 17 questions with a recall of 7 days. Each question has 5 standardized answer options with a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. A positive change from baseline indicates an improvement. Change from baseline in KOOS Function in daily living score was analyzed using a mixed effects model for repeated measures (MMRM) including all time-points to compare treatment groups. The model includes baseline, treatment, timepoint and treatment-by-timepoints as fixed effects. Missing data is assumed to be Missing at Random (MAR). Based on second secondary estimand framework.
Time Frame: Baseline, Weeks 1 (Day 5), 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | QUC398 300 mg | Placebo
Number analyzed (Participants) | 45 | 49
score on scale
  Week 1 (Day 5) | 2.9 (2.32) | 4.4 (2.22)
  Week 4: number analyzed (Participants) | 43 | 48
  Week 4 | 3.5 (2.33) | 10.5 (2.23)
  Week 8: number analyzed (Participants) | 41 | 44
  Week 8 | 9.4 (2.35) | 16.4 (2.26)
  Week 12: number analyzed (Participants) | 43 | 44
  Week 12 | 11.3 (2.34) | 19.1 (2.26)
  Week 16: number analyzed (Participants) | 43 | 47
  Week 16 | 12.5 (2.34) | 20.5 (2.25)
  Week 20: number analyzed (Participants) | 41 | 45
  Week 20 | 15.0 (2.36) | 20.6 (2.27)
  Week 24: number analyzed (Participants) | 38 | 45
  Week 24 | 13.5 (2.4) | 20.6 (2.28)
  Week 28: number analyzed (Participants) | 37 | 44
  Week 28 | 13.1 (2.43) | 21.9 (2.29)
  Week 32: number analyzed (Participants) | 36 | 44
  Week 32 | 13.4 (2.46) | 21.7 (2.3)
  Week 36: number analyzed (Participants) | 33 | 37
  Week 36 | 14.3 (2.52) | 23.2 (2.39)
  Week 40: number analyzed (Participants) | 29 | 29
  Week 40 | 17.0 (2.62) | 22.5 (2.55)
  Week 44: number analyzed (Participants) | 26 | 27
  Week 44 | 16.3 (2.72) | 19.7 (2.66)
  Week 48: number analyzed (Participants) | 23 | 23
  Week 48 | 15.8 (2.85) | 25.4 (2.83)
  Week 52: number analyzed (Participants) | 25 | 23
  Week 52 | 16.4 (2.87) | 24.2 (2.91)

8. Secondary Outcome: Change From Baseline in Knee Injury and Osteoarthritis Outcome Score (KOOS) Function in Sport and Recreation Subscale
Description: The KOOS questionnaire is a commonly used instrument to assess the patient's perception about their knee and associated problems. The original KOOS consists of 5 subscales. One of those is the function in sport and recreation consisting of 5 questions with a recall of 7 days. Each question has 5 standardized answer options with a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. A positive change from baseline indicates an improvement. Change from baseline in KOOS Function in sport and recreation score was analyzed using a mixed effects model for repeated measures (MMRM) including all time-points to compare treatment groups. The model includes baseline, treatment, timepoint and treatment-by-timepoints as fixed effects. Missing data is assumed to be Missing at Random (MAR). Based on second secondary estimand framework.
Time Frame: Baseline, Weeks 1 (Day 5), 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | QUC398 300 mg | Placebo
Number analyzed (Participants) | 45 | 49
score on scale
  Week 1 (Day 5) | 2.1 (2.76) | 2.5 (2.65)
  Week 4: number analyzed (Participants) | 43 | 48
  Week 4 | 4.5 (2.78) | 7.5 (2.65)
  Week 8: number analyzed (Participants) | 41 | 44
  Week 8 | 8.7 (2.81) | 11.5 (2.7)
  Week 12: number analyzed (Participants) | 43 | 44
  Week 12 | 10.1 (2.79) | 17.3 (2.7)
  Week 16: number analyzed (Participants) | 43 | 47
  Week 16 | 12.0 (2.79) | 15.8 (2.67)
  Week 20: number analyzed (Participants) | 41 | 45
  Week 20 | 11.1 (2.82) | 16.7 (2.7)
  Week 24: number analyzed (Participants) | 38 | 45
  Week 24 | 12.6 (2.87) | 22.0 (2.71)
  Week 28: number analyzed (Participants) | 37 | 44
  Week 28 | 12.2 (2.9) | 19.4 (2.73)
  Week 32: number analyzed (Participants) | 36 | 44
  Week 32 | 14.2 (2.93) | 21.2 (2.74)
  Week 36: number analyzed (Participants) | 33 | 37
  Week 36 | 14.6 (3.00) | 22.1 (2.86)
  Week 40: number analyzed (Participants) | 29 | 29
  Week 40 | 12.4 (3.13) | 19.8 (3.06)
  Week 44: number analyzed (Participants) | 26 | 27
  Week 44 | 14.4 (3.25) | 22.5 (3.17)
  Week 48: number analyzed (Participants) | 23 | 23
  Week 48 | 12.9 (3.4) | 24.1 (3.36)
  Week 52: number analyzed (Participants) | 25 | 23
  Week 52 | 14.7 (3.42) | 23.2 (3.47)

9. Secondary Outcome: Change From Baseline in Knee Injury and Osteoarthritis Outcome Score (KOOS) Knee Related Quality of Life Subscale
Description: The KOOS questionnaire is a commonly used instrument to assess the patient's perception about their knee and associated problems. The original KOOS consists of 5 subscales. One of those is the knee-related quality of life consisting of 4 questions with a recall of 7 days. Each question has 5 standardized answer options with a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. A positive change from baseline indicates an improvement. Change from baseline in KOOS Knee related quality of life score was analyzed using a mixed effects model for repeated measures (MMRM) including all time-points to compare treatment groups. The model includes baseline, treatment, timepoint and treatment-by-timepoints as fixed effects. Missing data is assumed to be Missing at Random (MAR). Based on second secondary estimand framework.
Time Frame: Baseline, Weeks 1 (Day 5), 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | QUC398 300 mg | Placebo
Number analyzed (Participants) | 45 | 49
score on scale
  Week 1 (Day 5) | 0.4 (2.28) | 5.2 (2.2)
  Week 4: number analyzed (Participants) | 43 | 48
  Week 4 | 2.2 (2.3) | 5.7 (2.21)
  Week 8: number analyzed (Participants) | 41 | 44
  Week 8 | 5.3 (2.32) | 8.6 (2.24)
  Week 12: number analyzed (Participants) | 43 | 44
  Week 12 | 5.5 (2.31) | 11.5 (2.24)
  Week 16: number analyzed (Participants) | 43 | 47
  Week 16 | 8.6 (2.31) | 12.9 (2.22)
  Week 20: number analyzed (Participants) | 41 | 45
  Week 20 | 8.4 (2.33) | 12.3 (2.24)
  Week 24: number analyzed (Participants) | 38 | 45
  Week 24 | 7.1 (2.37) | 13.4 (2.25)
  Week 28: number analyzed (Participants) | 37 | 44
  Week 28 | 9.8 (2.39) | 16.3 (2.27)
  Week 32: number analyzed (Participants) | 36 | 44
  Week 32 | 9.5 (2.42) | 13.1 (2.28)
  Week 36: number analyzed (Participants) | 33 | 37
  Week 36 | 9.4 (2.48) | 15.8 (2.36)
  Week 40: number analyzed (Participants) | 29 | 29
  Week 40 | 10.4 (2.58) | 17.4 (2.52)
  Week 44: number analyzed (Participants) | 26 | 27
  Week 44 | 9.5 (2.68) | 16.7 (2.62)
  Week 48: number analyzed (Participants) | 23 | 23
  Week 48 | 11.1 (2.8) | 19.5 (2.77)
  Week 52: number analyzed (Participants) | 25 | 23
  Week 52 | 13.1 (2.79) | 17.6 (2.81)

10. Secondary Outcome: Change From Baseline in Patient's Global Assessment (PGA) as Assessed by NRS
Description: The PGA of osteoarthritis disease activity was performed using a NRS (11-point scale from 0 - 10) with a recall period of 24 hours, and it was completed by the participant prior to drug administration at visits specified in the assessment schedule. A negative change from baseline implied improvement in pain. Change from baseline in function in patients global assessment (PGA) was analyzed using a MMRM including all time-points to compare treatment group. The model included baseline, treatment, timepoint and treatment-by-timepoints as fixed effects. Missing data is assumed to be Missing At Random (MAR). Based on second secondary estimand framework.
Time Frame: Baseline, Weeks 1 (Day 5), 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | QUC398 300 mg | Placebo
Number analyzed (Participants) | 45 | 49
score on scale
  Week 1 (Day 5) | -0.1 (0.14) | -0.4 (0.13)
  Week 4: number analyzed (Participants) | 43 | 48
  Week 4 | -0.3 (0.2) | -0.8 (0.19)
  Week 8: number analyzed (Participants) | 41 | 44
  Week 8 | -0.7 (0.22) | -1.2 (0.21)
  Week 12: number analyzed (Participants) | 42 | 44
  Week 12 | -1.0 (0.27) | -1.4 (0.26)
  Week 16: number analyzed (Participants) | 42 | 47
  Week 16 | -1.0 (0.27) | -1.6 (0.26)
  Week 20: number analyzed (Participants) | 40 | 44
  Week 20 | -1.0 (0.30) | -1.7 (0.29)
  Week 24: number analyzed (Participants) | 37 | 45
  Week 24 | -1.2 (0.32) | -1.8 (0.3)
  Week 28: number analyzed (Participants) | 35 | 43
  Week 28 | -1.3 (0.33) | -2.1 (0.31)
  Week 32: number analyzed (Participants) | 36 | 43
  Week 32 | -1.3 (0.35) | -2.0 (0.33)
  Week 36: number analyzed (Participants) | 32 | 36
  Week 36 | -1.3 (0.33) | -2.3 (0.31)
  Week 40: number analyzed (Participants) | 27 | 27
  Week 40 | -1.4 (0.39) | -2.1 (0.38)
  Week 44: number analyzed (Participants) | 23 | 25
  Week 44 | -1.5 (0.38) | -2.2 (0.37)
  Week 48: number analyzed (Participants) | 22 | 22
  Week 48 | -1.3 (0.42) | -2.3 (0.41)
  Week 52: number analyzed (Participants) | 24 | 21
  Week 52 | -1.5 (0.47) | -2.0 (0.47)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus follow up period, up to a maximum duration of approximately 60 weeks.
Groups:
- Total: Total
Arm/Group | QUC398 300 mg | Placebo | Total
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/51 | 0/101
Serious Adverse Events (participants affected / at risk) | 2/50 | 4/51 | 6/101
Other Adverse Events (participants affected / at risk) | 41/50 | 37/51 | 78/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QUC398 300 mg (N=50) | Placebo (N=51) | Total (N=101)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 1
Chest pain (General disorders) | 0 | 1 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Syncope (Nervous system disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QUC398 300 mg (N=50) | Placebo (N=51) | Total (N=101)
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 3
Influenza like illness (General disorders) | 8 | 4 | 12
Injection site reaction (General disorders) | 23 | 5 | 28
COVID-19 (Infections and infestations) | 4 | 2 | 6
Influenza (Infections and infestations) | 6 | 10 | 16
Nasopharyngitis (Infections and infestations) | 7 | 11 | 18
Pneumonia (Infections and infestations) | 1 | 3 | 4
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 4
Urinary tract infection (Infections and infestations) | 0 | 3 | 3
Muscle strain (Injury, poisoning and procedural complications) | 0 | 3 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 10 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 0 | 5
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 10 | 2 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3 | 4
Synovial cyst (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3
Headache (Nervous system disorders) | 4 | 3 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 5

LIMITATIONS AND CAVEATS:
The decision to terminate the study early, resulted in fewer participants contributing data at the later timepoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-11-28): https://cdn.clinicaltrials.gov/large-docs/90/NCT05462990/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-23): https://cdn.clinicaltrials.gov/large-docs/90/NCT05462990/SAP_001.pdf